CLINICAL TRIAL: NCT06579625
Title: The Effect of Health Belief Model-Based Cancer Education Given to Caregivers of Cancer Patients on Cancer Information Load, Knowledge and Attitudes Towards Cancer Screenings
Brief Title: The Effect of Health Belief Model-Based Cancer Education on Cancer Information Load, Knowledge and Attitudes Towards Cancer Screenings
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Semanur AKER, nurse, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AnkaraU-HEM-SA-01
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Cancer; Education; Caregiver; Randomised Controlled Trial
Keywords: Cancer; Cancer Screening; Caregiver; Health Belief Model; Information; Attitude; Health Education
MeSH Terms: conditions — Neoplasms; Behavior; Health Education

STUDY DESIGN:
Intervention Model Description: two group with a of Health Belief Model-Based cancer education control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Other): The effect of cancer education on cancer knowledge burden, information about cancer screenings, and attitudes will be evaluated by providing cancer education to 39 patients in the experimental group.
  Interventions: Other: Cancer education
- Control group (No Intervention): The control group will not receive any intervention.

INTERVENTIONS:
Other: Cancer education — Participants in the experimental group will receive cancer education.
  Arms: experimental group

SUMMARY:
Participants will be randomly assigned to the experimental and control groups. The study will involve a total of 78 participants, with 39 in the experimental group and 39 in the control group. The 39 participants assigned to the experimental group will first complete the cancer knowledge burden, and attitudes and information about cancer screenings scales. They will then receive cancer education consisting of four modules, which will be completed over four weeks. At the end of these four weeks, they will complete the scales again. One month after the education, the experimental group will complete the scales once more for follow-up monitoring. The control group will first complete the cancer knowledge burden, and attitudes and information about cancer screenings scales after agreeing to participate in the study. They will complete the scales again one month later. The evaluation of the education in the experimental group will involve comparing the scales completed before and after the education.

DETAILED DESCRIPTION:
Cancer is a significant public health issue with high morbidity and mortality rates worldwide and in our country. According to cancer statistics published by the World Health Organization's International Agency for Research on Cancer, the number of people diagnosed with cancer increases every year. In 2022, the global number of new cancer cases was 20 million, and it is estimated to reach 32.6 million by 2045. Cancer ranks second among all causes of death globally and in Turkey, with approximately one in every six individuals succumbing to cancer according to WHO estimates. The increasing number of cancer cases day by day unders cores the importance of cancer as it exerts physical, emotional, and financial pressure on individuals, families, and society and is a significant cause of death.

In secondary prevention methods for cancer prevention, early diagnosis and screening programs encompass the diagnosis and treatment of the disease before it progresses. In our country, cancer screenings include breast cancer, cervical cancer, and colon cancer screenings. It is important to raise awareness in the community about early diagnosis and screening programs for cancer. All individuals in the society should learn the causes, risk factors, and symptoms of cancer from accurate and reliable sources. Research results indicate that participants knowledge about cancer screenings is not at a sufficient level. With the high prevalence of cancer in society, individuals are increasingly seeking information about cancer. However, as knowledge about cancer increases, individuals may experience information overload, which can lead to confusion. Studies have shown that as the burden of cancer knowledge increases, individuals tend to avoid cancer-related information and engage in fewer health-protective, preventive behaviors.

The Health Belief Model pos its that individuals health behaviors are influenced by beliefs, values, and attitudes and is frequently used in health education. The primary aim of the Health Belief Model is to understand what motivates individuals to engage in preventive behaviors, to undergo health screenings forearly diagnosis, and to control the in diseases, and to develop interventions tailored to the individual. This study aims to evaluate the effect of cancer educati on based on the Health Belief Model on the knowled geand attitudes towards cancer screenings among caregivers of cancer patients.

The population of the study consists of individual sproviding care to cancer patients who have agreed to participate in the research, aged between 30 and 70 years, literate, and with out anyyisual, auditory, intellectual, or orthopedic impairments. Th eincluded individuals (78 caregivers) will be stratified by the clinics where they provide care and weighted according to the number of inpatients they carefor. The experimental and control groups will be listed and numbered separately for each clinic, and random sampling will be conducted using a real random number generator (https://www.random.org/). Random selections will be planned sequentially, with one experimental and one control group alternately. Selection will continue until the sample size is reached. As part of thepre-test, the introductory information form, Cancer Knowledge Scale, Cancer Screening Knowledge Scale, and Cancer Screening Attitude Scale will be administered to individuals in both the experimental and control groups. The experimental group will receive a 4-week cancer education program based on the Health Belief Model, while no interventi on will be made for the control group. As part of the post-test, the Cancer Knowledge Scale, Cancer Screening Knowledge Scale, and Cancer Screening Attitude Scale will be administered to both the experimental and control groups. Data analysis will be performed using the Statistical Package for Social Sciences (SPSS) 25.0 program.

Cancer screenings ensure the early detection of cancer. Cancers diagnosed in the early stages are easier, faster, and more cost-effective to cure and treat compared to advanced-stage cancers. This study may provide guid an ceto caregivers of cancer patients by increasing their knowledge about cancer and cancer screening programs, reducing the burden of cancer knowledge, and increasing participation rates in screenin gprograms. Additionally, this study may shed light on the impact of cancer education on cancer knowledge, screening knowledge, and attitudes among individuals with different demographic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who agree to participate in the study, are aged 30-70,
* Are literate,
* Do not have any auditory, visual, cognitive, or orthopedic disabilities that would prevent participation,
* Are not receiving palliative care services, will be included. This includes caregivers of cancer patients.

Exclusion Criteria:

* Individuals under the age of 30 or over the age of 70,
* Those who are illiterate,
* Those with disabilities that would prevent participation in the study,
* Those who provide care for cancer patients receiving palliative care services will not be included in the study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-10-28 (Estimated)

PRIMARY OUTCOMES:
İnformation Towards Cancer Screening Scale | one month
  The scale consists of 15 items and is unidimensional. It is a five-point Likert scale. The items on the scale are answered on a range from 1 to 5 as follows: "5: Strongly agree, 4: Agree, 3: Neither agree nor disagree, 2: Disagree, 1: Strongly disagree."
  The scale is suitable for use with men and women aged 30-70 who are at least literate and do not have cognitive, visual, or orthopedic disabilities that would prevent them from answering the scale. The administration method of the scale should be such that the researcher observes the participant, and the participant reads and answers the scale items independently. The scale can be used in any situation where it is necessary to measure attitudes towards cancer screenings, provided that the appropriate sample and administration method are used.
  The lowest possible score on the scale is 15 and the highest is 75. There is no specific cutoff point for the scale. Scores close to 15 indicate

SECONDARY OUTCOMES:
Cancer Knowledge Burden | one month
  Cancer information overload was measured using a thirteen- item battery assessing feelings about the overwhelming quantity of cancer information. Four response options (strongly disagree to strongly agree) were provided for each item (i.e., higher scores for greater overload). Items were crafted based on HINTS questions, an explication of the construct (detailed in the literature review of this article), and formative research conducted by the authors.
Attitudes Towards Cancer Screening Scale | one mounth
  The scale consists of 24 items and is unidimensional. It is a five-point Likert scale. The items on the scale are answered on a range from 1 to 5 as follows: "5: Strongly agree, 4: Agree, 3: Neither agree nor disagree, 2: Disagree, 1: Strongly disagree."
  The scale is suitable for use with men and women aged 30-70 who are at least literate and do not have cognitive, visual, or orthopedic disabilities that would prevent them from answering the scale. The administration method of the scale should be such that the researcher observes the participant, and the participant reads and answers the scale items independently. The scale can be used in any situation where it is necessary to measure attitudes towards cancer screenings, provided that the appropriate sample and administration method are used.
  The lowest possible score on the scale is 24 and the highest is 120. There is no specific cutoff point for the scale. Scores close to 24 indicat

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abdurrhman Yurtaslan Oncology Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No